CLINICAL TRIAL: NCT01268449
Title: Phase 1 Evaluation of Low Dose Laser in Treatment of Tinnitus
Brief Title: Evaluation of Low Dose Laser in Treatment of Tinnitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Islamic Azad University of Mashhad (Other)
Responsible Party: Dr. Mahboobeh Adami Dehkordi, Islamic Azad University Mashad Branch
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Laser-tinnitus-202
Record Dates: First submitted 2010-12-29; First posted 2010-12-30 (Estimated); Last update posted 2010-12-30 (Estimated); Status verified 2010-08

CONDITIONS: Subjective Tinnitus
Keywords: Tinnitus; Low power laser
MeSH Terms: conditions — Tinnitus | interventions — Lasers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Laser group (Active Comparator)
  Interventions: Radiation: Low dose laser
- Placebo group (Placebo Comparator): Randomly,half of the patients receive placebo.
  Interventions: Radiation: Placebo

INTERVENTIONS:
Radiation: Low dose laser — 5mv laser with a wavelength of 650nm
  Arms: Laser group
Radiation: Placebo — The act of radiating laser to the ear is done while the set is off.
  Arms: Placebo group

SUMMARY:
The purpose of this study is to determine wether low dose laser is effective on idiopathic subjective tinnitus.

ELIGIBILITY:
Inclusion Criteria:

* Adults older than 18 years old
* Idiopathic, subjective, unilateral tinnitus with at least 2 month duration

Exclusion Criteria:

* Patients with chronic otitis media
* Patients with tympan perforation with any underlying cause
* Patients with external otitis
* Patients with tinnitus related to a retrocochlear lesion or other known lesions of the ear

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2008-03; Primary Completion 2010-08 (Actual); Study Completion 2010-09 (Actual)